CLINICAL TRIAL: NCT00320684
Title: A Positron Emission Tomography Study of the Serotonin Transporter in Weight-Restored Women With Anorexia Nervosa
Brief Title: Serotonin Transporter Concentrations in Women With a History of Anorexia Nervosa
Status: Completed | Type: Observational
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: #4625/5767R; K23MH002021 (NIH); DATR AK-TNNS1
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Eating Disorders; Anorexia Nervosa
Keywords: Serotonin Transporter; Positron-Emission Tomography
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Women who have had anorexia nervosa but are now maintaining a healthy weight
- 2: Women who have never had anorexia nervosa and are maintaining a healthy weight

SUMMARY:
This study will compare the concentrations of serotonin transporter in the brains of women with a history of anorexia nervosa who are currently maintaining a normal weight to those of healthy women of normal weight.

DETAILED DESCRIPTION:
Anorexia nervosa (AN) is a serious eating disorder that is associated with substantial morbidity and mortality. Despite being dangerously underweight, people with AN believe that they are overweight, and frequently exhibit symptoms of depression and anxiety. Other symptoms of AN include the following: resistance to maintaining a healthy body weight; fear of gaining weight or becoming overweight; and denial of the seriousness of one's current low body weight. Relapse rates for AN are extremely high. Serotonin is a neurotransmitter, or chemical messenger, that affects mood, impulse control, and appetite. A serotonin transporter is a specialized protein that allows cells to communicate with each other by using serotonin. Disturbances in the serotonergic system, the network of nerve cells that uses serotonin as its neurotransmitter, may contribute to the behaviors that are characteristic of AN. This study will compare women with a history of AN who are now maintaining a normal weight to healthy women of normal weight in terms of the concentration of serotonin transporter in their brains.

Participants in this observational study will undergo one positron emission tomography (PET) scan and one magnetic resonance imaging (MRI) scan. Both will be used to measure the concentration of the serotonin transporter. A radioactive tracer will be used for the PET scan, and will be administered via an intravenous catheter line. No treatment will be provided in this study.

ELIGIBILITY:
Inclusion Criteria:

* History of anorexia nervosa
* BMI has been greater than 18.5 kg/m² for at least 9 months
* Agrees to use an effective method of contraception
* Off all psychotropic and other types of medications likely to impact the serotonin system for at least 21 days

Exclusion Criteria:

* Use of any psychotropic medication or other types of medications that are likely to affect the serotonin system within 21 days of study entry
* Current DSM-IV Axis-I diagnosis of any illness other than an eating disorder
* Current AN or history of AN within 9 months prior to study entry
* Presence of any psychiatric symptom that would make participation unsafe
* Significant active physical illnesses, particularly those that may affect the brain or serotonergic system, including the following: blood dyscrasias lymphomas; hypersplenism; endocrinopathies; renal failure or chronic obstructive lung disease; autonomic neuropathies; low hemoglobin; anemia; peripheral vascular disease; and malignancy
* Currently receiving effective medication treatment for an eating disorder
* History of Raynaud's phenomena and/or acrocyanosis
* Significant regular tobacco use (defined as more than 1 pack per week)
* Lacks capacity to consent
* Pregnant
* Breastfeeding
* Any metal implants, pacemaker, metal prostheses, orthodontic appliances, or the presence of shrapnel
* Significant history of claustrophobia that would complicate the completion of MRI
* Current or past radiation exposure in the workplace or as part of a research protocol in the previous year
* Badged for radiation

Inclusion for Healthy Controls:

* Female age 18-45
* BMI >18.5 kg/m
* Drug and medication free
* Willingness to engage in effective birth controls

Exclusion for Healthy Controls

* History of any DSM-IV Axis - I diagnosis
* History of Axis II disorder that would be accompanied by impulse control problems or significant suicidal behavior
* Significant active physical illness
* Lacks capacity to consent
* Pregnancy, currently lactating
* Metal implants, pacemaker or metal prostheses or orthodontic appliances or shrapnel
* Current, past radiation exposure in the workplace or as part of a research protocol in the previous year or badged for radiation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be women who have recovered from anorexia nervosa and are currently living in the local community.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2003-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn Attia, MD, Principal Investigator — New York State Psyciatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- See also: Click here for the New York State Psychiatric Institute Eating Disorders Clinic website — http://www.columbiaeatingdisorders.org